CLINICAL TRIAL: NCT05917691
Title: Impact of Functional Status on 30-day Resource Utilization and Organ System Complications Following Index Bariatric Surgery: a Cohort Study
Brief Title: Impact of Functional Status on 30-day Resource Utilization and Organ System Complications Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Zhiyi Zuo, MD, Principal Investigator, University of Virginia
Other Study IDs: HSRZOKZZ2
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Dependence; Perioperative/Postoperative Complications; Frailty
MeSH Terms: conditions — Postoperative Complications; Frailty | interventions — Bariatric Surgery; Anesthetics, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dependent functional status: 223 patients; "dependent" for those documented as "partially dependent" or "totally dependent."
  Interventions: Procedure: Bariatric surgery; Drug: General anesthetic; Device: Indeterminate
- Independent functional status: 65404 patients; "independent" for those documented as such.
  Interventions: Procedure: Bariatric surgery; Drug: General anesthetic; Device: Indeterminate

INTERVENTIONS:
Procedure: Bariatric surgery — Current Procedural Terminology (CPT) codes: 43644, 43645, 43770, 43775, 43842, 43843, 43845, 43846, 43847.
Drug: General anesthetic — Cases were required to have a documented "general anesthesia" anesthetic technique. Administered drugs were otherwise indeterminate under the current study design (observational study of a deidentified database).
Device: Indeterminate — Devices were indeterminate under the current study design (observational study of a deidentified database).

SUMMARY:
The goal of this observational study is to assess the effect of functional status on bariatric surgical thirty-day outcomes. The main questions it aims to answer are:

* Is functional status associated with higher incidence of 30-day unplanned resource utilization?
* Is functional status associated with higher incidences of secondary adverse events?

Participants will be sampled from the 2015-2019 American College of Surgeons National Surgical Quality Improvement Program

ELIGIBILITY:
Inclusion Criteria:

* Current Procedural Terminology (CPT) codes: 43644, 43645, 43770, 43775, 43842, 43843, 43845, 43846, 43847
* Elective, non-emergent cases
* "General surgery" surgical specialty
* "General anesthesia" anesthetic technique

Exclusion Criteria:

* Documented concurrent or other procedures
* Patients admitted to the hospital for greater than one day preceding surgery
* Acute kidney injury (preoperative)
* End-stage renal disease (preoperative)
* Metastatic disease (preoperative)
* Wound infection (preoperative)
* Sepsis (preoperative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elective bariatric surgical patients, ACS-NSQIP 2015-2019
Sampling Method: Non-Probability Sample
Enrollment: 65627 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Unplanned resource utilization (composite) | 30 days
  A composite binary outcome comprising unplanned readmission, return to the operating room, or prolonged (≥ 30 day) length of stay.

SECONDARY OUTCOMES:
Composite organ system complications | 30 days
  Cardiac complications included cardiac arrest and myocardial infarction. The only neurologic complication that was captured was stroke/cerebrovascular accident. Respiratory complications included reintubation, prolonged ventilatory wean, and pneumonia. Hematologic/infectious complications included superficial surgical site infection (SSI), deep incisional SSI, organ space SSI, wound dehiscence, bleeding, sepsis, septic shock, deep venous thrombosis, and pulmonary embolism. Renal complications included progressive renal insufficiency and acute kidney injury.
Mortality | 30 days
  Mortality

IPD SHARING:
Plan to Share IPD: Yes
American College of Surgeons National Surgical Quality Improvement Program and the hospitals participating in the ACS NSQIP are the source of the data used herein. The Participant Use Data File (PUF) is a Health Insurance Portability and Accountability Act (HIPAA)-compliant data file containing cases submitted to the American College of Surgeons National Surgical Quality Improvement Program®. To request a copy of the PUF, individuals (data recipients) must agree to comply with the terms and conditions set forth in the Data Use Agreement, provide contact information, and complete a short online questionnaire. Once the information provided by the data recipient is received and processed by ACS NSQIP staff, a website address will be submitted electronically to the data recipient. The data recipient will then have 10 days (240 hours) to visit the website and download the data file.

REFERENCES:
- Available data/document: Individual Participant Data Set — https://www.facs.org/quality-programs/data-and-registries/acs-nsqip/participant-use-data-file/